CLINICAL TRIAL: NCT01520129
Title: Pilot Study of Interpersonal and Social Rhythm Therapy for Subthreshold Bipolar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Holly Swartz, Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11110666
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Bipolar Disorder NOS
Keywords: Bipolar Disorder; Bipolar NOS; Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interpersonal and social rhythm therapy (Other): IPSRT Subjects will receive weekly 45 minute sessions of IPSRT for 20 weeks. IPSRT sessions focus on reducing symptoms by teaching patients to: a) increase regularity of social rhythms and regulate sleep-wake cycles; b) resolve interpersonal problems that contribute to mood symptoms (role dispute, role transition, grief, or interpersonal deficits); and c) recognize and accept the symptoms of subthreshold BP disorder (psychoeducation). Although we train therapists in techniques that are specific to each component, in practice, these strategies are administered flexibly and fluidly, without distinct boundaries between modalities. During the course of a session, therapists move seamlessly among the techniques, according to patients' needs.
  Interventions: Other: Interpersonal and social rhythm therapy

INTERVENTIONS:
Other: Interpersonal and social rhythm therapy — IPSRT Subjects will receive weekly 45 minute sessions of IPSRT for 20 weeks. IPSRT sessions focus on reducing symptoms by teaching patients to: a) increase regularity of social rhythms and regulate sleep-wake cycles; b) resolve interpersonal problems that contribute to mood symptoms (role dispute, role transition, grief, or interpersonal deficits); and c) recognize and accept the symptoms of subthreshold BP disorder (psychoeducation). Although we train therapists in techniques that are specific to each component, in practice, these strategies are administered flexibly and fluidly, without distinct boundaries between modalities. During the course of a session, therapists move seamlessly among the techniques, according to patients' needs.
  Other Names: IPSRT

SUMMARY:
The investigators propose to conduct a 20 week open pilot study of Interpersonal and Social Rhythm Therapy (IPSRT) to treat individuals (n=18) with subthreshold bipolar (BP) who are currently depressed. The investigators will conduct a preliminary evaluation of sleep-wake and social rhythm patterns in study participants using questionnaires and actigraphy. Primary aims of this study are to evaluate feasibility of this treatment and assessment approach. Exploratory aims are to examine 1) sleep-wake and social rhythm patterns in subthreshold BP, 2) impact of IPSRT on symptoms and functioning over time and 3) relationship between sleep-wake and social rhythm patterns and treatment outcomes.

DETAILED DESCRIPTION:
Subthreshold bipolar disorder (BP) is a common, understudied, illness associated with high levels of impairment. "Subthreshold" BP refers to individuals who have episodes of both depression and hypomania, but the episodes of hypomania do not last long enough or are characterized by too few symptoms to meet conventional criteria for "threshold" hypomania. Compared to individuals with episodes of depression only (major depressive disorder or MDD), individuals with subthreshold BP have higher rates of suicide, earlier onset of illness, more episodes of depression, and more co-occurring psychiatric disorders. Despite the severity of the disorder, virtually nothing is known about how to treat this illness.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 - 65
2. Meets criteria for bipolar disorder NOS, currently in an episode of major depression, as defined by the DSM-IV (American Psychiatric Association, 1994) and documented by the use of the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I), and by a rating of >15 on the 25-item Hamilton Rating Scale for Depression (HRSD-25). We will limit inclusion specifically to those individuals who have histories of 1) at least one short (2-3 day) hypomanic episode OR 2) at least one subthreshold hypomanic episode (at least 4 consecutive days of elevated mood and 2 of the other symptoms of hypomania or irritable mood with 3 of the other symptoms of hypomania). NOTE: Like the National Comorbidity Survey Replication, individuals whose hypomania occurred while on antidepressant medication will not be excluded from the trial (Merikangas, personal communication, 2011).
3. Ability and willingness to give informed, written consent.
4. Subjects may participate in this study if they are currently taking psychotropic medications at time of informed consent. They will start study interventions if they still meet eligibility criteria after a one week wash-out period.
5. Ability and willingness to participate in study procedures

Exclusion Criteria:

1. Severe or poorly controlled concurrent medical disorders that may cause confounding depressive symptoms (i.e., untreated hypothyroidism or lupus) or require medication(s) that could cause depressive symptoms (i.e., high doses of beta blockers or alpha interferon)
2. Meets criteria for one of the following concurrent DSM-IV psychiatric disorders: any psychotic or organic mental disorder, bipolar I disorder, bipolar II disorder, current alcohol or drug dependence, primary obsessive compulsive disorder or primary eating disorders. (primary refers to the diagnosis associated with the most functional impairment); borderline personality disorder; antisocial personality disorder
3. Acute suicidal or homicidal ideation or requiring psychiatric hospitalization. Subjects who require inpatient treatment will be excluded (or discontinued) from the study and referred to one of WPIC's inpatient mood disorder units, or, if preferred, to an inpatient facility nearer to the patient's home
4. Severe cognitive deficits that would preclude treatment with psychotherapy and/or prevent completion of study questionnaires
5. Non-fluent in English. Subjects must be able to speak and understand English because one of the study interventions, IPSRT, is an experimental talk-therapy. The DMDPP does not have multilingual therapists.
6. Current participation in another form of individual psychotherapy. Concurrent participation in couples therapy, peer support groups (such as Alcoholics Anonymous), or family therapy will be permitted
7. Prior lack of response to a trial of at least 12 weeks of IPSRT conducted by a qualified IPSRT therapist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Depression severity | 20 weeks
  The primary endpoint is depression severity at week 20, which will be measured via the Hamilton Rating Scale for Depression 25-item score (HRSD-25) and the Young Mania Rating Scale (YMRS).

CONTACTS AND LOCATIONS:
Overall Officials: Holly Swartz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Depression and Manic Depression Prevention Program, Pittsburgh, Pennsylvania, United States